CLINICAL TRIAL: NCT04728763
Title: Aspergillosis and Humoral Alveolar Immunity by Proteomics
Acronym: ASPEOMIC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201003
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Aspergillus Fumigatus Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients for whom bronchial endoscopy with BAL is performed as part of an exploration of invasive pulmonary aspergillosis (IPA) or Chronic pulmonary aspergillosis (CPA) in current care :
  * Probable or proven invasive pulmonary aspergillosis according to the criteria of the EORTC (2019) or
  * Chronic pulmonary aspergillosis according to the criteria of ESCMID / ERS (2016)
  Interventions: Other: Protein profile
- Control Group: Patients for whom bronchial endoscopy with BAL is performed as part of an exploration of diffuse interstitial lung disease or a lower respiratory infection other than Aspergillus in routine care
  Interventions: Other: Protein profile

INTERVENTIONS:
Other: Protein profile — Analysis of the protein content by proteomics of bronchoalveolar lavage

SUMMARY:
Aspergillus fumigatus is the most common opportunistic mold found in lung fungal infections in humans. Aspergillus is the cause of invasive pulmonary aspergillosis with a poor prognosis in immunocompromised patients and the chronic pulmonary aspergillosis which affects 3 million patients worldwide, with underlying pulmonary pathologies such as tuberculosis and its sequelae. The medicinal means to fight against these different forms are limited and not very effective. In addition, the emergence of resistance makes the search for new therapeutic strategies of major importance.

The interaction between the fungal spore and our innate immune system is the first step leading to infection.

The innate immune system is made up of cellular immunity and humoral immunity. While the first is well described, the second, consisting of soluble mediators, is essential for anti-aspergillus immunity but relatively little studied. The study of soluble mediators present in the alveolar fluid interacting directly with the Aspergillus spore would make it possible to analyze the first stages of infection. The analysis of the proteome present in the bronchoalveolar lavage of uninfected patients, suffering from various forms of aspergillosis and suffering from other types of infections would make it possible to highlight the essential and specific components of anti- immunity aspergillary.

The objective of this study is to analyze the protein profiles of innate immunity in the pulmonary alveoli in the absence or presence of Aspergillus or non-fungal infection in order to highlight the soluble mediators of the more specific immunity of the Aspergillosis.

ELIGIBILITY:
Inclusion Criteria for the case group (IPA / CPA): :

1. Patient who are more than 18 years old
2. Patients for whom bronchial endoscopy with BAL is performed as part of an exploration of IPA or CPA in current care. Probable or proven invasive pulmonary aspergillosis according to the criteria of the EORTC (2019).
3. Patient who has given his consent.

Inclusion Criteria In the control group :

1. Patient who are more than 18 years old
2. Patients for whom bronchial endoscopy with BAL is performed as part of an exploration of diffuse interstitial lung disease or a lower respiratory infection other than Aspergillus in routine care. Chronic pulmonary aspergillosis according to the criteria of ESCMID / ERS (2016)
3. Patient who has given his consent.

Exclusion Criteria for the case and the control group:

1. Pregnant woman
2. Patient deprived of their rights
3. Patient under tutorship or guardianship or under the protection of a conservator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with or without pulmonary aspergillosis for whom a bronchial fibroscopy with bronchoalveolar lavage is performed as part of their care path.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Protein profile | at day 90
  Protein profiles of innate immunity in the pulmonary alveoli

IPD SHARING:
Plan to Share IPD: Undecided